CLINICAL TRIAL: NCT05936125
Title: Short Term Outcomes Of Tricuspid Valve Annuloplasty Using A Flexible Band
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Sayed, M.D. Mahmoud Kamel Mohamed Sayed, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 282
Record Dates: First submitted 2023-04-22; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Valvular Heart Disease; Tricuspid Valve Regurgitation
Keywords: Tricuspid Valve; Tricuspid Valve Regurgitation; Tricuspid Valve Annuloplasty
MeSH Terms: conditions — Heart Valve Diseases; Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with tricuspid valve regurgitation undergoing open heart surgery (Experimental): Patients undergoing open heart surgery (for any reason) with concomitant tricuspid valve regurgitation
  Interventions: Other: Annuloplasty Using Flexible Band

INTERVENTIONS:
Other: Annuloplasty Using Flexible Band — Tricuspid valve annuloplasty using a flexible band; (Polyethylene terephthalate band): (Dacron band)

SUMMARY:
Functional tricuspid regurgitation (FTR) remains a common finding in patients with left-sided valvular heart diseases especially mitral valve regurgitation or stenosis. It is mainly caused by dilatation and flattening of the tricuspid valve (TV) annulus as a result of right ventricular (RV) enlargement and is inevitably affected by the RV function. Multiple studies support the better outcome of using rigid ring annuloplasty over suture repair for treating FTR in concern with the durability and freedom from residual regurgitation. These studies refer the superiority of rigid ring annloplasty to the three-dimensional configuration achieved by such rings which matches the normal tricuspid annulus and, at the same time, to the rigid support of the annulus. On the other hand, other studies support the use of flexible prosthetic bands like Dacron or polytetrafluroethilin (PTFE), especially over suture techniques, due to their easy applicability and availability with good postoperative results. Therefore, suture annyloplasty became nowadays less convenient for FTR repair since both flexible bands and rigid rings appeared to offer good midterm outcomes in recent meta-analysis studies. However, the ideal annuloplasty method for repairing FTR is still debatable between the three-dimensional (3D) rigid rings versus flexible prosthetic bands. In this retrospective comparative study, we share our experience with flexible fashioned bands in FTR.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented at Assiut University Hospital with tricuspid valve regurgitation

Exclusion Criteria:

* Age less than 18 years old.
* Tricuspid valve stenosis.
* Organic tricuspid valve disease.
* Infective endocarditis on tricuspid valve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Tricuspid valve regurgitation | 1 year post operative
  Using Echocardiography to asset tricuspid valve regurgitation

SECONDARY OUTCOMES:
Tricuspid Annular Plane Systolic Excursion (TAPSE) | 1 year post operative
  Using Echocardiography to asset Tricuspid Annular Plane Systolic Excursion (TAPSE)

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Hospital University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided